CLINICAL TRIAL: NCT03510780
Title: Periodontal Regeneration With Platelet-rich Fibrin (Prf) and Autogenous Bone Graft (Abg) Versus Enamel Matrix Derivative (Emd) and Abg in the Treatment of Intrabony Periodontal Defects a Longitudinal Randomized Control Clinical Study
Brief Title: Platelet-rich Fibrin and Autogenous Bone vs Enamel Matrix Derivative and Autogenous Bone in Intrabony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, professor and chairman, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24042018
Record Dates: First submitted 2018-04-24; First posted 2018-04-27 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Periodontal Bone Loss; Periodontal Attachment Loss
Keywords: Platlet rich fibrin; Enamel Matrix Derivative; Bone graft; Non-inferiority study
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Attachment Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMD treated patients (Active Comparator): Periodontal surgery with Enamel Matrix Derivative is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. Autogenous corticocancellous BG material will be collected using bone scrapers EMD will be applied to the entire root surfaces ; then, ABG will be applied alternatively with EMD into the IBD according to the "sandwich" technique until the IBD will be completely filled. Finally the flap will be repositionated and sutures completed by interrupted sutures.
  Interventions: Procedure: Periodontal surgery with Enamel Matrix Derivative
- PRF treated patients (Experimental): Periodontal surgery with Platelet Rich Fibrin is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. Autogenous corticocancellous BG material will be collected using bone scrapers , the PRF membrane cut into small pieces and mixed with the ABG will be placed within the IBDs until they will be completely filled. Then the other two PRF membranes in each patient will be adapted over the grafted defect Finally horizontal mattress and interrupted sutures will be carried out.
  Interventions: Procedure: Periodontal surgery with Platlet Rich fibrin

INTERVENTIONS:
Procedure: Periodontal surgery with Enamel Matrix Derivative — Patients will be treated by periodontal surgical flaps with the addition of EMD + bone graft
  Arms: EMD treated patients
Procedure: Periodontal surgery with Platlet Rich fibrin — Patients will be treated by periodontal surgical flaps with the addition of PRF + bone graft
  Arms: PRF treated patients

SUMMARY:
Currently, the most positive documented outcomes of periodontal regenerative therapy (PRT) in intrabony defects (IBDs) have been achieved with a combination of bone grafts ( BGs) and a regeneration material like membranes in guided tissue regeneration ( GTR) or enamel matrix derivative (EMD) in Induced Periodontal Regeneration ( IPR) technique. Among the graft materials only autogenous bone grafts ( ABGs).and demineralized freeze-dried bone allografts (DFDBA), are considered regenerative materials.

Polypeptide growth factors revealed a potential application in PRT periodontal because are the biological mediators during wound healing and regeneration and autologous platelet concentrates ( PC) constitute a safe and convenient approach to deliver them.

Among PC, platelet-rich fibrin ( PRF) belongs to a group of second-generation blood autologous products prepared by peripheral blood centrifugation without any nonclotting agent, so to obtain a dense three-dimensional clot architecture that concentrates platelets, fibrin, leukocytes, cytokines, and sustain cellular migration. This clot is then compressed to obtain elastic and very strong membranes that can be used directly as membranes or as a ﬁlling agent, after chopping, alone or in combination with BGs.

Several studies demonstrate that PRF is effective in promoting bone regeneration (BR) when used alone or in combination with BG during oral/ periodontal surgery.

To date, there are very few published clinical controlled trials that compare the results of PRF + BGs to the outcomes of PRF / BG alone in the treatment of IBDs and no study about PRF + ABG in the same defects. Only one case report tested the use of PRF + ABG mixed with bovine hydroxyapatite in the treatment of insufficient alveolar ridge width in aesthetic area. The aim of the present study is to verify if the combined use of PRF + ABG in the management of IBDs may be a treatment modality clinically "not inferior" to that with EMD + ABG.

DETAILED DESCRIPTION:
Experimental Design. This is a prospective, randomized and controlled clinical trial designed to evaluate the clinical and radiographic outcomes 12 months after two treatment modalities of IBDs: PRF + ABG into defects in the test subjects( TS); EMD + ABG in the control subjects ( CS). The patients enrolled exhibit unfavourable IBDs and all experimental sites will be accessed with a simplified papilla preservation flap ( SPPF) procedure. The filling material (ABG) is common to both treatments: therefore, the investigation will focus on the addictive effect of PRF used in place of EMD. EMD is chosen as the active control ( AC) as it is currently considered as the biological "gold standard" agent for the treatment of IBDs.

A non-inferiority trial ( NIT) is designed to prove that using PRF instead of EMD could achieve a similar result, reducing the treatment's cost and allowing the clinicians to use autogenous material only.

An AC (comparator) is present, but the investigators do not include a third experimental arm, a group of IBDs treated using Open Flap Debridement ( OFD) alone, as it is widely accepted in NITs.

The estimate of the AC effect vs. placebo is assumed from a recent meta-analysis, by the Lower Bound of a 95% Confidence Interval ( CI) of the mean of EMD + ABG, while an OFD estimate from the corresponding 95% CI Lower Bound is adopted by Venezia (2004). The difference between estimates is set as the added benefit of the AC and as a ground for the assay sensitivity.

Study Population. 44 patients affected by moderate-to-severe chronic periodontitis, will be selected for the study. Each patient will participate in the study with a single experimental site. The participants will receive verbal and written information and they will sign a consent form approved by the Ethical Committee of the G. D'Annunzio University of Chieti - medical faculty. The study protocol is in accordance with the Declaration of Helsinki of 1975, revised in Tokyo in 2004. Four months before the surgical treatment, all 44 patients will undergo SRP by ultrasonic instruments and hand curettes and motivational instructions on oral home care.

Non-inferiority margin. A reliable estimate of the expected clinical attachment level ( CAL) gain from an EMD + ABG treatment is drawn from a recent meta-analysis, reporting on 548 IBDs in 434 patients.

The CAL Gain Median was M=3.76 (SD=1.07) with 95% . Prudently the CI Lower Bound (3.48 mm) is chosen as estimate of EMD + ABG CAL gain.

By literature, CAL gain obtainable by OFD surgical treatments alone is 2.47 mm. The differential effect of using EMD amounts about 1 mm.

In accordance with the 95% - 95% method (the Fixed Margin approach), a magnitude equal to the AC's expected effect (1 mm) is chosen for the M1 margin, to guarantee the new treatment's efficacy. For clinical relevance, a second M2 margin is prefigured to preserve at least a further 50% (0.5 mm) of the comparator's effect. Both M1 and M2 will be adopted for the secondary outcomes.

Sample Size and Randomization. Not knowing a priori whether the collected data will meet the assumptions and the conditions making sensible an analysis of covariance (ANCOVA), the sample size will be initially calculated for an analysis of variance (ANOVA).

With one-tail , an α == 0.05, a power 1-β = = 0.90 and a SD = = 1.07 mm 1, a sample size of 20 patients per group is needed to detect the margin M1 = 1 mm in CAL gain between the groups.

Assuming that it will became possible to conduct an ANCOVA, the sample size sufficient to detect an M2 margin will be calculated. If to detect a ∆M1=1 mm with ANOVA a total sample size of N=40 will be required, adjusting for baseline values allowed to halve the margin (∆M2=0.5) adding only 2 more patients.

Each defect will be assigned a defect number and will be randomly allocated to one of the two treatment regimens. Assignment will be performed by a custom made computer-generated table. To conceal allocation, opaque envelopes will be assigned to the specific experimental site and will be opened during surgery.

Clinical Measurements.Complete oral and periodontal examinations will be performed for each patient 3 months after SRP. These included FMPS, FMBS, PPD, CAL, and gingival recession ( GR) for six sites per tooth (mesiobuccal, mid-buccal, disto-buccal, mesio-lingual/ palatal, mid-lingual/palatal, and disto-lingual/palatal sites). Clinical measurements at experimental sites will be recorded using a University of North Carolina (UNC-15, HuFriedy, Chicago, Illinois, USA) periodontal probe. The measurements will be taken immediately before surgical treatment (baseline) and 1 year after treatment, by the same experienced examiner, who will be masked to the treatment..

Radiographic Measurements. Preoperative and 3- 6- 12-months postoperative intraoral standardized radiographs will be taken by the paralleling technique using an individual film-holder device consisting of a bite block rigidly connected to an acrylic dental splint to achieve identical film placement at each evaluation. Pre- and postoperative radiographs will be evaluated by two experienced clinicians who will be masked with respect to the provenience of the radiographs and the clinical measurements. The positions of alveolar crest level and of the bottom of the defect distance and will be marked by a pencil on the radiographs and bottom of the defect will be measured by a millimeter grid. Linear distances between the most coronal interproximal alveolar crest level and the bottom of the defect will be obtained by counting the grids.

Surgical Technique. All the surgeries will be performed by the same experienced clinician. Both in TS and CS, after local anaesthesia, mucoperiosteal SPPFs will be raised. The flap will be extended to the teeth mesial and distal to the tooth to be treated and, if necessary, mesial and distal vertical releasing incisions will be performed to allow more visibility and defects accessibility. After flap elevation, vestibular flap mobility will be tested to ensure that primary closure of the wound could be achieved through tension -free suturing. The granulation tissue adherent to the alveolar bone will be removed to provide full access and visibility to the root and bone surfaces; SRP will be performed, but no osseous recontouring. Autogenous corticocancellous BG material will be collected using bone scrapers in both the TS and CS adjacent areas.

Then, root surfaces in the CS will be conditioned for 2 minutes with 24% ethylenediaminetetraacetic acid (EDTA) and then thoroughly rinsed with saline solution. Before EMD application, single internal mattress suture at the defect- associated interdental area to reach primary closure of the papilla in the absence of any tension will be prepared by 4-0 sutures and left loose to apply EMD and the ABG. EMD will be applied to the entire root surfaces of the CS as well as to the alveolar bone; then, ABG will be applied alternatively with EMD into the IBD according to the "sandwich" technique until the IBD will be completely filled. Finally the flap will be repositioned and sutures completed by interrupted sutures.

In the TS, after the defect debridement, the PRF membrane cut into small pieces and mixed with the ABG will be placed within the IBDs until they will be completely filled. Then the other two PRF membranes in each patient will be adapted over the grafted defect extending over the periphery of the defect in the buccal and lingual directions in order to cover all the graft and recontour the bone architecture. Finally the flap will be repositioned and horizontal mattress and interrupted sutures will be carried out.

Data Processing. Since direct comparisons about single outcomes is the trial's scope, a multiple univariate analysis is chosen.

The primary outcome of the study is CAL gain at 12 months. Changes in PPD, GR and bottom of the defect distance are secondary outcomes.

Relying on previous studies and literature reporting a ρ between baseline- and gain-score in the order of 0.7. an ANCOVA (on gain scores with baseline scores as covariate) is designed as the main analysis. Furthermore, by virtue of the expected correlation, sample size could be reduced to ¼.

Nonetheless, an ANOVA is performed as well, both for comparison and as a reference in sample size calculation.

Non-inferiority is assessed by mean of CI of the main outcome's gain-scores difference between the two treatments. For the non-inferiority to be established, the CI Upper Bound should neither touch nor overrun the margin. Secondary outcomes will be analyzed similarly.

ELIGIBILITY:
Inclusion Criteria:

* a full-mouth plaque score (FMPS) 25 and a full-mouth bleeding score (FMBS) 26 < 20% at the time of surgery
* to have at least 20 teeth,; at least 1 tooth exhibiting vertical bone loss detected by radiographic examination (alveolar crest level [ ACL] - bottom of the defect [ BD] distance = Bone defect depth [ BDD]) ≥ 4 mm and a probing pocket depth (PPD) ≥ 5mm when evaluated 12 weeks after phase I non- surgical therapy [ scaling and root planing ( SRP)].

Exclusion Criteria:

* no systemic diseases
* no medications affecting periodontal status during the previous 6 months
* not pregnant or lactating; non-smoker
* and no periodontal therapy in the 2 previous years, no inadequate endodontic treatment, no dental mobility,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-07-02 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Periodontal attachment gain | 1 year
  Reduction of the distance between the cementum-enamel junction and the depth of the probable site

SECONDARY OUTCOMES:
Bone gain | 1 year
  Gain of bone into the periodontal defects

CONTACTS AND LOCATIONS:
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: Undecided